CLINICAL TRIAL: NCT03448172
Title: A Phase 1, Open Label, Single-period, Non-randomized Study To Evaluate The Pharmacokinetics, Excretion, Mass Balance, And Metabolism Of [14c]Pf-05221304 Administered Orally To Healthy Adult Male Subjects
Brief Title: Single-dose Study of [14C]PF-05221304 Metabolism and Excretion in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C1171010
Record Dates: First submitted 2018-02-07; First posted 2018-02-27 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Product (Experimental): [14C]PF-05221304
  Interventions: Drug: [14C]PF-05221304

INTERVENTIONS:
Drug: [14C]PF-05221304 — a single oral dose of [14C]PF-05221304 (50 mg/100 µCi liquid formulation)

SUMMARY:
The purpose of the study is to characterize the absorption, distribution, metabolism, and excretion (ADME) of a single oral dose of [14C]PF-05221304 in Healthy Adult Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Ages of 18 and 45 years, inclusive.
2. Body mass index (BMI) of >= 17.5 and <= 30.4 kg/m2
3. Total body weight > 50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, allergic disease or clinical findings.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Mass Balance | 0-96 hr
  Cumulative recovery of urinary, fecal, and total excretion of radioactivity over time expressed as percentage of total radioactive dose administered

SECONDARY OUTCOMES:
Metabolic profiling for PF-05221304 in plasma, urine, and feces | 0-96 hr
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces
Radioactivity AUClast | 0-96 hr
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for radioactivity
Plasma PF-05221304 AUClast | 0-96 hr
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-05221304
Radioactivity AUCinf | 0-96 hr
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for radioactivity
Plasma PF-05221304 AUCinf | 0-96 hr
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-05221304
Radioactivity Cmax | 0-96 hr
  Maximum Observed Plasma Concentration (Cmax) for radioactivity
Plasma PF-05221304 Cmax | 0-96 hr
  Maximum Observed Plasma Concentration (Cmax) for PF-05221304
Radioactivity Tmax | 0-96 hr
  Time to Reach Maximum Observed Plasma Concentration for radioactivity
Plasma PF-05221304 Tmax | 0-96 hr
  Time to Reach Maximum Observed Plasma Concentration for PF-05221304
Radioactivity t1/2 | 0-96 hr
  Plasma Decay Half-Life (t1/2) for radioactivity
Plasma PF-05221304 t1/2 | 0-96 hr
  Plasma Decay Half-Life (t1/2) for PF-05221304
Number of subjects experiencing an adverse event | Up to 28 days post dosing of IP on Day 1
  Assessment by physical examinations, adverse event monitoring, clinical laboratory measurements, vital signs and ECG.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity. Treatment-emergent are events between dosing with study drug and up to 28 days after that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171010&StudyName=A+Phase+1%2C+Open+Label%2C+Single-period%2C+Non-randomized+Study+To+Evaluate+The+Pharmacokinetics%2C+Excretion%2C+Mass+Balance%2C+And+Metabolism+Of+%5B14c%5Dpf-05221304+Administered+Orally+To+Healthy+Adult+Male+Subjects